Outcomes of small process groups on medical students' grit, resilience, and stress:

A quasi-experimental pilot study

Approved June 24, 2022

#### **Informed Consent**

(Introductory paragraph to the survey and Q1, informed consent):

You are invited to participate in a study of medical student wellbeing being conducted by the College of Osteopathic Medicine of the Pacific-NW.

You have been selected because you are a medical student at COMP-NW. [For the intervention group this will say: You have been selected because you are a medical student at COMP-NW and are participating in the small group sessions].

# **Overall Purpose of Study:**

This study is to assess measures of wellbeing for COMP-NW medical students from the beginning to the end of the year. These measures are important to be able to see if and how your wellbeing changes over time. From this information, we hope to be better able to assist and support you going forward.

#### **Explanation of Procedures:**

This survey should take about 15 minutes to complete. We are asking for your initials to be able to match your data up with the survey at the end of the year, but this will not be seen by anyone, and your data will be immediately de-identified in order to protect your answers. None of your answers will be shared as individual information or stored with your name. Your name and any identifying information will be removed from the data for any publication or presentation. [For intervention survey additional sentence: [The psychiatrist] will not know at any time if you are participating in the research study or not. At no time during the course of the academic year will [the psychiatrist] have access to your survey results.]

The second survey will be the same as this one. You will receive an email with the link at the end of the academic year. You are not required to take the second survey if you take this one, however this study uses pre/post data so your data may not be able to be used if you only take one survey. Therefore we encourage you to take both surveys.

### **Potential Risks and Discomforts:**

The survey questions ask you about certain things, like stress levels, that may cause some emotional discomfort if you are feeling stressed. You may stop the survey at any time, in which case your data will not be used. Please refer to the bottom of this form for information on resources the school offers for mental and emotional support.

## **Potential Benefits:**

Medical students are known to have higher levels of stress and anxiety than their peers. Studies like this one aim to find out more about what might help medical students with stress. By participating in this research you are providing information that may be used to develop programs and support resources for you and other medical students.

This section will only be in the intervention group survey:

### **Compensation for Participation:**

There will be a drawing of a \$100 gift card for students who participate in the full year of small group sessions].

### **Assurance of Confidentiality:**

Your initials will collected only to assign you an ID number and track your pre/post data, but will not be available to anyone except the primary researcher, who will never review the data with your initials attached. No identifying information about you will be used in any communications, presentations, or publications. The data you provide will be combined with other data in aggregate. Data and records created by this project are the property of the University and the investigator. You may have access to information collected on or about you by making a written request to the principal investigator. This right of access extends only to information collected on or about you and not to information collected on or about others participating in the project.

## **Statement of Injury or Special Costs:**

In the event that this research activity results in emotional or mental distress, you should contact the PI at [#] or [the psychiatrist] at [#]. Treatment will be available, including crisis care and follow-up care as needed. You and your third-party payer (such as health insurance) may need to provide payment for any such treatment. This paragraph does not mean that you are releasing or waiving any legal right you might otherwise have against the investigator or WESTERNU as a result of your participation in this research activity.

# Withdrawal from the Study:

Your participation is voluntary. Your decision whether or not to participate will not affect your present or future relationship with the university, college, or the researchers. If you decide to participate, you are free to withdraw your consent and to discontinue participation at any time up until submission for publication.

#### **Offer to Answer Questions:**

You should feel free to ask questions now or at any time during the study. If you have questions about this study, you can contact the PI at [email] or [#]. If you have questions about the rights of research subjects, contact the WESTERNU IRB Office, [#].

#### **Consent Statement:**

You are voluntarily making a decision whether or not to participate. Your selection of YES below indicates that you have decided to participate, having read the information provided above.

Q1: I have read this information, which is printed in English. This is a language that I read and understand.

[Survey multiple choice buttons: YES [directed to survey] NO ["Thank you." Directed out of survey.